CLINICAL TRIAL: NCT05498142
Title: Predicting the Risk of Venous Thromboembolism in Critically Ill Patients: Validation of Pre-existing Risk Prediction Models and Development of a Prediction Model
Brief Title: Predicting the Risk of Venous Thromboembolism in Critically Ill Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Frederik Keus, Principal Investigator, University Medical Center Groningen
Other Study IDs: VTEICU
Record Dates: First submitted 2022-08-09; First posted 2022-08-11 (Actual); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: Venous Thromboembolism; Critical Illness
MeSH Terms: conditions — Venous Thromboembolism; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- SICS I: Prospective cohort study based on the 'Simple Intensive Care Studies' (SICS) registry (NCT02912624)
- SICS II: Prospective cohort study based on the 'Simple Intensive Care Studies' (SICS) registry (NCT03577405)
- AFIB-ICU: An international inception cohort study.
- Emmen: Patients admitted to the ICU of a community hospital in the Netherlands.

SUMMARY:
Introduction: Venous thrombosis (VTE), including both deep vein thrombosis (DVT) and pulmonary embolism (PE) remains a frequent complication in patients admitted to the Intensive Care Unit (ICU). Multiple prediction models for estimating the risk of VTE have been developed. However, many models have not been externally validated. The aim of this study is to perform a comprehensive external validation of pre-existing prediction models for predicting the risk of in-hospital VTE in critically ill patients. In case current risk assessment models fail, the investigators aim to additionally develop and internally validate a new risk prediction model.

Methods: During the first phase of the study the investigators will perform external validation of existing prediction models. The performance, discrimination, calibration and clinical usefulness of the models will be evaluated. In the second phase of the study, in case performance of current risk assessment models is deemed insufficient for clinical application, the investigators will develop a model for predicting the risk of in-hospital VTE in critically ill patients. A multivariable prediction model will be constructed using a combination of predefined candidate predictors. This model will be internally validated and performance will be compared with performance of existing VTE risk prediction models.

Dissemination: This protocol will be published online. This study will be reported according to the Transparent reporting of a multivariable prediction model for individual prognosis or diagnosis (TRIPOD) statement and this study will be submitted to a peer-reviewed journal for publication.

DETAILED DESCRIPTION:
Objective

1. To perform external validation of existing prediction models (phase 1)
2. To develop and internally validate a model for predicting the risk of in-hospital VTE in critically ill patients (phase 2)

Study design:

The objectives will require a large number of outcome events (see sample size calculation). To fulfill this requirement and to increase generalizability of the results, the intention is to collect data from several sources, which will include several types of study designs. The investigators currently have access to data from the Simple Intensive Care studies' (SICS-I and SICS-II; clinicalTrials.gov identifier:NCT02912624 and NCT03577405). In addition, an unpublished database that contains registry data from a community-hospital in the Netherlands will be used. Third, data from the prospective AFIB-ICU cohort study will be used. To further increase the sample size, the investigators are exploring additional collaboration with colleagues aiming to include more data.

In the final manuscript a table with the following descriptives of each data source will be included: study design, selection criteria, time period of conduct; data collection (prospective, retrospective); and types and definitions of included predictor and outcome variables.

This study will be reported according to the Transparent reporting of a multivariable prediction model for individual prognosis or diagnosis (TRIPOD) statement.

Study participants:

The target population are critically ill patients who are admitted to the ICU regardless of underlying disease. Patients who were admitted after planned surgery or other procedures will be excluded. The investigators foresee that there will be differences between the selection criteria of each cohort. As stated above, the investigators will reflect on these differences in the final manuscript.

Candidate predictors:

Candidate predictors were selected based on the following criteria:

1. established or suggested association with VTE (based on literature)
2. or incorporation in another VTE risk assessment model;
3. and readily available and easy to obtain in daily clinical practice.

The following candidate predictors will be explored: active cancer, acute infection, acute renal failure, cardiovascular failure, central venous access, elderly age, estrogen therapy, sex, major surgery, mechanical ventilation, multiple trauma, obesity, previous VTE, reduced mobility, respiratory failure, stroke, thrombophilic disorder, vasopressor use. When available the investigators also aim to include C-reactive protein (CRP), hemoglobin (Hb), leukocytes and thrombocytes in the model. A complete list of all candidate predictors including their definitions and units of measurement, is displayed in table 1*.

Outcome:

The primary outcome will be in-hospital VTE. VTE will be defined as any objectively proven event occurring during initial hospital admission. No screening protocol will be used. DVT will include acute thrombosis of lower-extremity veins (iliac, femoral or popliteal), confirmed by compression ultrasonography, venography, CT, MRI, or autopsy. Pulmonary embolism will be defined as acute thrombosis within the pulmonary vasculature as shown by ventilation-perfusion scan, CT angiography, or autopsy. Upper extremity DVT will be included in the model but venous thrombosis in any other site (e.g. portal vein thrombosis) will be excluded as these may represent a different entity.

Data management:

Data from multiple cohorts will be collected and stored in a secure location in any applicable format in compliance with institutional, national and international applicable regulatory laws.

Identifying and inclusion of previous risk assessment models:

A recently published systematic review will be used to select the prediction models for external validation6. Additionally, the investigators will contact experts in the field and conduct a non-structured literature search to identify any additional and/or more recently published prediction models for in-hospital VTE. The following online libraries will be searched: Embase, Medline and Google Scholar. No time restrictions will be used. Models will be selected for inclusion if all predictor variables are available.

Sample size:

For the two phases of this study: external validation of existing prediction models and, second, development and internal validation of a new model for predicting the risk of in-hospital VTE in critically ill patients, the required sample size will be calculated in two different ways.

Phase 1: external validation of existing prediction models The investigators will assess whether the collected data are sufficient for external validation by calculating the sample size for external validation according to a recently published study. For each risk assessment model, a sample size calculation will be performed.

Phase 2: development and internal validation of a model for predicting the risk of in-hospital VTE in critically ill patient In phase 2, the sample size needed to develop and internally validate the model was calculated according to a recently published method for sample size calculation for prediction models. Sample size calculation was based on a binary prognostic outcome, the estimated area under the curve (AUC), the estimated amount of candidate prognostic variables and the estimated outcome proportion. An AUC of 0.75 was used as baseline. Assuming an outcome prevalence of 3% in the study sample implicates that apporoximately 7600 patients need to be included to register 230 events for the evaluation of 22 candidate predictor variables.

Statistical analysis:

All analyses will be conducted after data collection has been completed according to, and after publishing of, this protocol. Deviations from this protocol will be reported accordingly in the final manuscript. Patient characteristics will be presented as means (with standard deviations; SD) or medians (with interquartile ranges; IQR) depending on distributions. Categorical data will be presented as proportions. Where appropriate, the investigators will account for clustering between cohorts from different sources independently using meta-analytic techniques.

External validation of existing prediction models:

For external validation, the overall model predictive performance, calibration, discrimination and clinical usefulness will be tested. Overall predictive performance will be tested using Nagelkerke's R2. Discrimination, which is the ability to distinguish patients with and without VTE, will be quantified using the concordance (C) statistic, identical to the area under the curve in a receiver operating characteristic curve. Calibration, which is the agreement between predicted and observed frequency, will be evaluated by modeling a regression line with intercept (α) and slope (β). Decision curve analysis will be performed to evaluate clinical usefulness of prediction models compared to alternative strategies (such as 'treat all patients' or 'treat no patients').

Development and internal validation of a prediction model:

This second objective will only be pursued if external validation of existing models appears insufficient for clinical use and if the predefined effective sample size has been reached. A multivariable prediction model for estimating VTE risk will be constructed. Subsequently, the score will be internally validated to correct for optimism. Normality of the data will be assessed using P-P plots and histograms. Linearity will be assessed using scatter plots. Differences between continuous variables will be assessed using Student's t-tests or Mann-Whitney-U test where appropriate.

The model will be constructed using the following steps:

1. Candidate predictor selection criteria were described above. Definitions are displayed in table 1*.
2. Missing variables (<25%) will be imputed using multiple imputations. Missing variables (>25%) will be excluded. Multiple imputations for missing outcome data will not be performed and patients with missing VTE data will be excluded from all analyses.
3. A binary logistic regression model will be constructed using in-hospital VTE as dependent outcome and the candidate predictors as independent variables. Continuous variables will not be converted to categorical variables. The aim is to include as few variables as reasonably possible to increase simplicity and enhance clinical applicability. Variables will be included based on previous knowledge, clinical reasoning, and observed strengths of associations. The investigators will not use a prespecified significance threshold for elimination. Results will be presented as adjusted Odds ratios (OR) with 95% confidence intervals (CI) and regression coefficients (β-values).
4. The logistic model will be converted to a clinically usable risk assessment model using methods previously described in the Framingham Heart Study. Additionally, the full model will be presented.
5. Internal validation will be performed using bootstrapping
6. Several tests for evaluation of model performance will be used. Overall predictive performance will be tested using Nagelkerke's R2. Discrimination, which is the ability to distinguish patients with and without VTE, will be quantified using the concordance statistic (C). Calibration is by definition expected to be good in the development cohort, and this will be assessed by modeling a regression line with intercept (α) and slope (β). The apparent and optimism-corrected model performance estimates will both be presented.

Data management and analysis will be conducted using STATA version 14.0 or newer (StataCorp, College Station, TX) or R software.

Ethics:

Patients gave informed consent for participation in the SICS-I and SICS-II studies (METc M15.168207). For the registry database a waiver for informed consent was provided (METc M11.104639 and M16.193856). For the AFIB ICU study informed consent from patients or surrogates will be obtained if needed as per national laws.

*Tables 1 is available upon request, please refer to the primary investigator.

ELIGIBILITY:
Inclusion Criteria:

1. Emergency admission

   Exclusion Criteria:
2. Age < 18 years
3. Planned admission either after surgery or for other reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population are critically ill patients who are admitted to the ICU regardless of underlying disease. We will exclude patients who were admitted after planned surgery or other procedures. We foresee that there will be differences between the selection criteria of each cohort. We will reflect on these differences in the final manuscript
Sampling Method: Probability Sample
Enrollment: 7600 (Estimated)
Dates: Start 2015-03 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Number of patients with in-hospital VTE | Initial hospital admission
  VTE will be defined as any objectively proven event occurring during initial hospital admission. No screening protocol will be used. DVT will include acute thrombosis of lower-extremity veins (iliac, femoral or popliteal), confirmed by compression ultrasonography, venography, CT, MRI, or autopsy. Pulmonary embolism will be defined as acute thrombosis within the pulmonary vasculature as shown by ventilation-perfusion scan, CT angiography, or autopsy. We will include upper extremity DVT in the model but exclude venous thrombosis in any other site (e.g., portal vein thrombosis) as these may represent a different entity.

REFERENCES:
- [Background] Wetterslev M, Moller MH, Granholm A, Haase N, Hassager C, Lange T, Hastbacka J, Wilkman E, Myatra SN, Shen J, An Y, Siegemund M, Young PJ, Aslam TN, Szczeklik W, Aneman A, Arabi YM, Cronhjort M, Keus F, Perner A. New-onset atrial fibrillation in the intensive care unit: Protocol for an international inception cohort study (AFIB-ICU). Acta Anaesthesiol Scand. 2021 Jul;65(6):846-851. doi: 10.1111/aas.13827. Epub 2021 Apr 23. PMID 33864378
- [Background] Gaus H, Gulzow M, Meyer-Hofmann G. [Late lesions following thorotrast use]. Klin Wochenschr. 1966 Jan 1;44(1):32-9. doi: 10.1007/BF01747176. No abstract available. German. PMID 5984857
- [Background] Spyropoulos AC. Upper vs. lower extremity deep vein thrombosis: outcome definitions of venous thromboembolism for clinical predictor rules or risk factor analyses in hospitalized patients. J Thromb Haemost. 2009 Jun;7(6):1041-2. doi: 10.1111/j.1538-7836.2009.03351.x. No abstract available. PMID 19548912
- [Background] Darzi AJ, Repp AB, Spencer FA, Morsi RZ, Charide R, Etxeandia-Ikobaltzeta I, Bauer KA, Burnett AE, Cushman M, Dentali F, Kahn SR, Rezende SM, Zakai NA, Agarwal A, Karam SG, Lotfi T, Wiercioch W, Waziry R, Iorio A, Akl EA, Schunemann HJ. Risk-assessment models for VTE and bleeding in hospitalized medical patients: an overview of systematic reviews. Blood Adv. 2020 Oct 13;4(19):4929-4944. doi: 10.1182/bloodadvances.2020002482. PMID 33049056
- [Background] Riley RD, Debray TPA, Collins GS, Archer L, Ensor J, van Smeden M, Snell KIE. Minimum sample size for external validation of a clinical prediction model with a binary outcome. Stat Med. 2021 Aug 30;40(19):4230-4251. doi: 10.1002/sim.9025. Epub 2021 May 24. PMID 34031906
- [Background] Riley RD, Ensor J, Snell KIE, Harrell FE Jr, Martin GP, Reitsma JB, Moons KGM, Collins G, van Smeden M. Calculating the sample size required for developing a clinical prediction model. BMJ. 2020 Mar 18;368:m441. doi: 10.1136/bmj.m441. No abstract available. PMID 32188600
- [Background] Van Calster B, Nieboer D, Vergouwe Y, De Cock B, Pencina MJ, Steyerberg EW. A calibration hierarchy for risk models was defined: from utopia to empirical data. J Clin Epidemiol. 2016 Jun;74:167-76. doi: 10.1016/j.jclinepi.2015.12.005. Epub 2016 Jan 6. PMID 26772608
- [Background] Vickers AJ, Elkin EB. Decision curve analysis: a novel method for evaluating prediction models. Med Decis Making. 2006 Nov-Dec;26(6):565-74. doi: 10.1177/0272989X06295361. PMID 17099194
- [Background] Janssen KJ, Donders AR, Harrell FE Jr, Vergouwe Y, Chen Q, Grobbee DE, Moons KG. Missing covariate data in medical research: to impute is better than to ignore. J Clin Epidemiol. 2010 Jul;63(7):721-7. doi: 10.1016/j.jclinepi.2009.12.008. Epub 2010 Mar 24. PMID 20338724
- [Background] Sullivan LM, Massaro JM, D'Agostino RB Sr. Presentation of multivariate data for clinical use: The Framingham Study risk score functions. Stat Med. 2004 May 30;23(10):1631-60. doi: 10.1002/sim.1742. PMID 15122742
- [Background] Viarasilpa T, Panyavachiraporn N, Marashi SM, Van Harn M, Kowalski RG, Mayer SA. Prediction of Symptomatic Venous Thromboembolism in Critically Ill Patients: The ICU-Venous Thromboembolism Score. Crit Care Med. 2020 Jun;48(6):e470-e479. doi: 10.1097/CCM.0000000000004306. PMID 32187076
- [Background] Schunemann HJ, Cushman M, Burnett AE, Kahn SR, Beyer-Westendorf J, Spencer FA, Rezende SM, Zakai NA, Bauer KA, Dentali F, Lansing J, Balduzzi S, Darzi A, Morgano GP, Neumann I, Nieuwlaat R, Yepes-Nunez JJ, Zhang Y, Wiercioch W. American Society of Hematology 2018 guidelines for management of venous thromboembolism: prophylaxis for hospitalized and nonhospitalized medical patients. Blood Adv. 2018 Nov 27;2(22):3198-3225. doi: 10.1182/bloodadvances.2018022954. PMID 30482763